CLINICAL TRIAL: NCT06284213
Title: Biomarkers for Vascular Contributions to Cognitive Impairment and Dementia Consortium
Acronym: MarkVCID
Status: Active, not recruiting | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Duke University (Other); Johns Hopkins University (Other); University of New Mexico (Other); University of Southern California (Other); University of Kentucky (Other); Rush University Medical Center (Other); University of Maryland, Baltimore (Other); University of California, San Francisco (Other); University of California, Los Angeles (Other); University of California, Davis (Other); University of Texas (Other); The University of Texas Health Science Center at San Antonio (Other); The University of Texas Health Science Center, Houston (Other); Mayo Clinic (Other); University of Mississippi Medical Center (Other); Washington University School of Medicine (Other); Olive View-UCLA Education & Research Institute (Other)
Responsible Party: Principal Investigator, Steven M. Greenberg, MD,PhD, Director, Hemorrhagic Stroke Research, Massachusetts General Hospital
Other Study IDs: 5U24NS100591 (NIH)
Record Dates: First submitted 2024-02-16; First posted 2024-02-28 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Cognitive Impairment; Dementia
Keywords: Biomarkers
MeSH Terms: conditions — Cognitive Dysfunction; Dementia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The MarkVCID study will collect serum, plasma, and packed cell samples from all participants each year, as possible. Consortium sites are expected to collect and store for consortium use between 4-5ml plasma, 4-5ml serum (5ml preferred for both sample types when possible), and 3-4ml packed cells for DNA extraction.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Normal Cognition (NC) with at least 1 vascular risk factor: NC is defined as:
  1. No diagnosis of SCD, MCI, or dementia; AND
  2. CDR: Sum of Boxes = 0 AND neuropsychological testing in normal range.
  Participants must have at least 1 of the following criteria prior to enrollment:
  Diabetes (at least 1):
  * Fasting (8-hour) blood sugar ≥126 mg/dL
  * Random or Post-prandial blood sugar ≥200 mg/dL
  * HbA1C ≥6.5%
  * Treatment with anti-diabetic medicine
  Hypertension plus (at least 2):
  * Use of anti-hypertensive medications for lowering blood pressure for ≥10 years
  * Current use of 2 or more anti-hypertensive meds for lowering blood pressure
  * Blood pressure in a research or clinical setting in the last 2 years with SBP ≥140 or DBP ≥90
  * Second blood pressure reading in a research or clinical setting in the last 2 years (different date) with SBP ≥140 or DBP ≥90
  * Evidence of likely HTN end organ damage
  MRI factors (at least 1):
  * Peri-Ventricular Fazekas Extent Grade or Deep Fazekas Extent Grade ≥2
  * ≥1 microbleeds
  * ≥1 lacunar infarcts
  Interventions: Other: No interventions
- Subjective Cognitive Decline (SCD): Subjective cognitive decline is defined as:
  1. Cognitive concerns based on a Short eCog-12 score ≥ 3 (based on administration to participant), AND
  2. Normal cognition (neuropsychological testing within normal range).
  Interventions: Other: No interventions
- Mild Cognitive Impairment (MCI): Mild cognitive impairment is defined as:
  1. There is a cognitive concern, i.e., the subject, the co-participant, or a clinician is concerned about a change in cognition compared to the subject's previous level.
  2. There is impairment in one or more cognitive domains (memory, language, executive function, attention, and visuospatial skills) that is greater than would be expected for the patient's age and educational background.
  3. There is largely preserved independence in functional abilities (no change from prior level of functioning or requires only extra effort and minimal aids or assistance).
  4. There is no evidence of dementia (cognitive changes are mild and there is no evidence of a significant impairment in social or occupational functioning).
  Interventions: Other: No interventions
- Mild Dementia: Mild dementia is defined as:
  1. The subject has cognitive or behavioral (neuropsychiatric) symptoms that meet all of the following criteria:
     1. Interfere with ability to function as before at work or at usual activities?
     2. Represent a decline from previous levels of functioning?
     3. Are not explained by delirium or major psychiatric disorder? AND
  2. Impairment in one* or more of the following domains.
     1. Impaired ability to acquire and remember new information.
     2. Impaired reasoning and handling of complex tasks, poor judgment.
     3. Impaired visuospatial abilities.
     4. Impaired language functions.
     5. Changes in personality, behavior, or comportment * In the event of single-domain impairment (e.g., language in PPA, behavior in bvFTD, posterior cortical atrophy), the subject must not fulfill criteria for MCI.
     AND
  3. CDR: Global Score = 0.5 or 1
  Interventions: Other: No interventions

INTERVENTIONS:
Other: No interventions — This is an observational study with no interventions.

SUMMARY:
Biomarkers for Vascular Contributions to Cognitive Impairment and Dementia (MarkVCID) is an NIH-funded consortium dedicated to finding biomarkers involved in age-related thinking and memory problems. Alzheimer's disease and other dementias leave signatures on brain scans or in the blood called biomarkers. The MarkVCID study will measure a panel of candidate biomarkers in 1800 participants and watch them closely to see what they tell us about changes in brain function and risk of memory loss.

Age-related problems in thinking and memory represent some of the greatest risks to public health in the US and globally. Diseases that affect small blood vessels in the brain have been shown to be major contributors to these changes. However, research and patient care can be held back by limited biomarkers that identify who should be treated.

The MarkVCID Consortium includes 17 US medical centers, a Coordinating Center, an External Advisory Committee, and NIH leadership. Data and biospecimens collected as part of this research study will be stored in a research database and biorepositories, so that researchers can use this information to study brain function.

DETAILED DESCRIPTION:
Biomarkers for Vascular Contributions to Cognitive Impairment and Dementia (MarkVCID) is an NIH-funded multisite consortium dedicated to developing promising predictive, diagnostic, target engagement and progression candidate biomarkers of small vessel disease in VCID. MarkVCID is a collaborative consortium of nine North American research sites (consisting of 17 institutions nationwide), a Coordinating Center, External Advisory Committee, and NIH leadership.

MGH serves as the Consortium's Coordinating Center and is comprised of an administrative and data core providing participating research sites with a common support infrastructure that facilitates cross-site collaborations, oversees development of standard operating procedures and data collection methods and manages consortium-wide data.

In phase two of the MarkVCID study, research sites are charged with enrolling and following ≥200 diverse human subjects with cognitive complaints and/or early symptomatic stages of cognitive impairment and dementia potentially associated with cerebrovascular small vessel disease. Sites will share data with the Coordinating Center which will be used for validation studies of chosen consortium biomarkers. Throughout the duration of the study, sites will utilize harmonized procedures and data collection methods to engage in multi-site biomarker validation. Both Cores comply with regulations for the protection of human research subjects (including Good Clinical Practices (GCP), 21 Code of Federal Regulations (CFR)) and with the International Conference on Harmonization (ICH) Regulations E2A and E6.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 60 and ≤ 90 years
* Diagnosis of normal cognition with at least one criterion for vascular risk*, subjective cognitive decline (preliminary diagnosis based on self-report question or eCog-12), mild cognitive impairment, or mild dementia based on standard research criteria
* Fluent in English or Spanish
* No contraindications to MRI including CVR
* No confounding neurologic, psychiatric, or medical disease

  *Participants with normal cognition must meet at least one criterion (diabetes, OR hypertension plus, OR MRI factors) for vascular risk prior to enrollment:
* Diabetes (at least one of the following):

  * Fasting (8-hour fast, usually overnight) blood sugar ≥126 mg/dL (≥7 mmol/L, or ≥1260 mg/L)
  * Random or Post-prandial blood sugar ≥200 mg/dL (≥11.11 mmol/L, or ≥2000 mg/L)
  * HbA1C ≥6.5% (or ≥47.5412 mmol/mol)
  * Treatment with an anti-diabetic medicine
* Hypertension plus (at least two of the following):

  * Use of anti-hypertensive medications for lowering blood pressure for ≥ 10 years
  * Current use of two or more anti-hypertensive medications for lowering blood pressure
  * One measured blood pressure in a research or clinical setting in the last 2 years with SBP ≥140 or DBP ≥90
  * A second measured blood pressure in a research or clinical setting on a different date in the last 2 years with SBP ≥140 or DBP ≥90
  * Evidence of likely HTN end-organ damage (e.g., LVH, albuminuria, eGFR<60, CHF)
* MRI factors (at least one of the following):

  * Peri-Ventricular Fazekas Extent Grade or Deep Fazekas Extent Grade ≥ 2
  * 1 or more microbleeds
  * 1 or more lacunar infarcts

Exclusion Criteria:

* Neurologic Disease: Based on the available data and investigator's impression, exclude those with confounding neurologic disease that would interfere with test performance or with biomarker analysis:

  * Frontotemporal lobar degeneration (FTLD)
  * Lewy body dementia (LBD)
  * Parkinson's disease
  * Multi system atrophy
  * Traumatic brain injury (TBI)-related cognitive impairment
  * TBI that interferes with MRI biomarker analyses (e.g., large volume traumatic lesion)
  * Non-small vessel strokes that interfere with test performance (e.g., post-stroke cognitive impairment or aphasia)
  * Non-small vessel strokes that interfere with MRI biomarker analysis (e.g., large volume strokes)
  * CADASIL (Cerebral Autosomal Dominant Arteriopathy with Subcortical Infarcts and Leukoencephalopathy)
  * Individuals known to be receiving, or planning to receive, anti-amyloid immunotherapy*
  * Other neurologic conditions that interfere with test performance or biomarker analysis

    * Individuals prescribed anti-amyloid immunotherapy after MarkVCID enrollment should be kept in the study.
* Medical and Psychiatric Conditions: Exclude those with medical and psychiatric conditions that would confound the course or interfere with test performance:

  * Schizophrenia or other active/severe psychotic disorders
  * Medical or psychiatric conditions likely to interfere with participation or retention (e.g., metastatic or malignant CNS cancer, active/severe depression or anxiety, HIV- Associated Neurocognitive Disorder)
  * Contraindications to MRI procedures, such as:

    * Claustrophobia
    * Cardiac pacemaker
    * Intracranial clips/metal implants
  * Contraindications to CVR:

    * COPD or other respiratory condition requiring oxygen therapy
    * Asthma or other respiratory condition requiring current use of medications such as inhalers

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will be selected from a variety of sources across the MarkVCID Consortium sites. These sources include, but are not limited to:
  * MarkVCID1 or other research studies
  * Alzheimer's Disease Research Center database
  * Patient registries such as Volunteer for Health
  * Community centers or organizations
  * Clinics:
    * Primary care
    * Neurology
    * Stroke Center
    * Outpatient Diabetes
    * Memory & Aging
Sampling Method: Non-Probability Sample
Enrollment: 1892 (Actual)
Dates: Start 2021-09-29 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
SVD progression as measured by decline in global cognition | The cognitive battery is implemented, and global cognition calculated, at Baseline and Years 1, 2 and 3 post-baseline.
  Global cognition scores will be calculated at each study timepoint as an average of age- and education-specific z-scores, based on tests scores from the MarkVCID2 cognitive battery (MoCA, Neuropsychological Testing Battery, Clinical Dementia Rating), which is based on Version 3 of the National Alzheimer's Coordinating Center's (NACC) Uniform Data Set (UDS) (Besser 2018).

SECONDARY OUTCOMES:
SVD progression as measured by decline in executive function | The cognitive battery is implemented, and executive function calculated, at Baseline and Years 1, 2 and 3 post-baseline.
  The measure of executive function is the Uniform Data Set (v3.0) executive function composite score (UDS3-EF) developed by Staffaroni et al (2021). The UDS3-EF is calculated from the following tests: Category Fluency - Animals; Verbal Fluency - Phonemic Tests (words beginning with F); Number Span Test (Backward); and Trail Making Tests A and B.

CONTACTS AND LOCATIONS:
Overall Officials: Steven M. Greenberg, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (17):
- United States (17):
  - University of Southern California, Los Angeles, California
  - University of California Los Angeles, Los Angeles, California
  - University of California Davis, Sacramento, California
  - University of California San Francisco, San Francisco, California
  - Olive View - UCLA Medical Center, Sylmar, California
  - Mayo Clinic Florida, Jacksonville, Florida
  - Rush University Medical Center & Illinois Institute of Technology, Chicago, Illinois
  - University of Kentucky, Lexington, Kentucky
  - University of Maryland, Baltimore, Baltimore, Maryland
  - Johns Hopkins University, Baltimore, Maryland
  - Mayo Clinic Rochester, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Washington University in St. Louis, St Louis, Missouri
  - University of New Mexico, Albuquerque, New Mexico
  - University of Texas Southwestern, Dallas, Texas
  - University of Texas Health Science Center Houston, Houston, Texas
  - University of Texas Health Science Center San Antonio, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Yes
MarkVCID research openly shares both within and outside the MarkVCID Consortium to the greatest extent practical. As per the MarkVCID Consortium's Charter, MarkVCID investigators are granted broad access to MarkVCID data, samples, analytic tools, and other resources with relevant permissions in place. MarkVCID data and samples may also be shared with external collaborators in compliance with the Consortium's external data sharing policies outlined in the MarkVCID Data Use Agreement. The process for requesting data and biosamples is described below.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Internal
  All MarkVCID research sites sign a Consortium Research Agreement governing the sharing of data and biosamples. Data entered in MarkVCID data systems by the research sites becomes available to all MarkVCID members, in accordance with the MarkVCID Data Sharing, Analysis, and Publications Policy and the MarkVCID Research Agreement.
  External
  If the request is approved by the MarkVCID Steering Committee, external users sign the DUA to gain access to the data. If biosamples are requested, external users will execute a Material Transfer Agreement (MTA) with the institution(s) providing samples. Biosamples typically ship within 3 months. Electronic data stored by the MarkVCID Consortium repository becomes available to the investigator about 3 weeks after project approval and signing of the DUA. Investigators requesting access to data and biosamples not held by the MarkVCID repository must contact relevant institution(s) and are subject to longer wait times.
Access Criteria: A MarkVCID Project Proposal Form must be submitted for data and biosample requests. The form requires an overview, a description of requested data and/or biosamples, assays, experiments to be conducted, and publication plans. Data requests will be reviewed by the Sharing Subcommittee and biosample requests by the Fluid-Based Biomarkers Subcommittee. Reviews will be based on scientific rationale, overlap with already approved analyses, and, for biosample requests, the scientific priority of the study relative to the number of available biosamples. The Steering Committee will then review proposal recommendations and determine approval. Investigators with approved proposals will sign a DUA and receive applicable data via Globus encrypted transfer. Investigators with approved biosample requests will execute necessary MTAs and receive deidentified biosamples from holding sites.
  Internal requests related to primary hypotheses of prespecified biomarker kits are exempt from the above.

REFERENCES:
- [Background] Besser L, Kukull W, Knopman DS, Chui H, Galasko D, Weintraub S, Jicha G, Carlsson C, Burns J, Quinn J, Sweet RA, Rascovsky K, Teylan M, Beekly D, Thomas G, Bollenbeck M, Monsell S, Mock C, Zhou XH, Thomas N, Robichaud E, Dean M, Hubbard J, Jacka M, Schwabe-Fry K, Wu J, Phelps C, Morris JC; Neuropsychology Work Group, Directors, and Clinical Core leaders of the National Institute on Aging-funded US Alzheimer's Disease Centers. Version 3 of the National Alzheimer's Coordinating Center's Uniform Data Set. Alzheimer Dis Assoc Disord. 2018 Oct-Dec;32(4):351-358. doi: 10.1097/WAD.0000000000000279. PMID 30376508
- [Background] Staffaroni AM, Asken BM, Casaletto KB, Fonseca C, You M, Rosen HJ, Boxer AL, Elahi FM, Kornak J, Mungas D, Kramer JH. Development and validation of the Uniform Data Set (v3.0) executive function composite score (UDS3-EF). Alzheimers Dement. 2021 Apr;17(4):574-583. doi: 10.1002/alz.12214. Epub 2020 Nov 20. PMID 33215852
- [Derived] Kern KC, Vohra M, Thirion ML, Wang DJJ, Wilcock DM, Thompson JF, Rosenberg GA, Sagare A, Moghekar A, Lu H, Lee T, Elahi FM, Satizabal CL, Tracy R, Seshadri S, Schwab K, Helmer K, Singh H, Kivisakk P, Greenberg SM, Vossel K, Kramer JH, Maillard P, DeCarli CS, Hinman JD. White matter free water mediates the associations between placental growth factor, white matter hyperintensities, and cognitive status. Alzheimers Dement. 2025 Feb;21(2):e14408. doi: 10.1002/alz.14408. Epub 2024 Dec 18. PMID 39692213